CLINICAL TRIAL: NCT01898585
Title: An Open-Label, Single-Arm, Multicenter Study To Assess The Safety Of Vemurafenib In Patients With Braf V600 Mutation Positive Metastatic Melanoma In South Africa.
Brief Title: An Open-Label Study of Zelboraf (Vemurafenib) in Patients With Braf V600 Mutation Positive Metastatic Melanoma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML28711
Record Dates: First submitted 2013-07-09; First posted 2013-07-12 (Estimated); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Malignant Melanoma
MeSH Terms: conditions — Melanoma | interventions — Vemurafenib

ARMS (1):
- Zelboraf Arm (Experimental)
  Interventions: Drug: Zelboraf

INTERVENTIONS:
Drug: Zelboraf — Vemurafenib 960 mg twice a day until progressive disease, unacceptable toxicity, consent withdrawal, death, reasons deemed by the treating physician or study termination.

SUMMARY:
This open-label, single-arm, multicenter study will assess the safety and efficacy of Zelboraf (vemurafenib) in patients with Braf V600 mutation positive metastatic melanoma. Patients will receive Zelboraf 960 mg twice a day until progressive disease, unacceptable toxicity, consent withdrawal, death, reasons deemed by the treating physician or study termination.

ELIGIBILITY:
Inclusion Criteria:

* Adults patients >= 18 years of age
* Patients with histologically confirmed metastatic melanoma (surgically incurable and unresectable stage IIIC or stage IV; AJCC) with documented BRAF V600 mutation determined by the cobas® BRAF V600 Mutation Test prior to administration of vemurafenib. Unresectable stage IIIC disease must have confirmation from a surgical oncologist
* Patients with either measurable or non-measurable disease (RECIST Version 1.1)
* Patients may or may not have received prior systemic therapy for metastatic melanoma
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2
* Patients must have recovered from all side effects of their most recent systemic or local treatment for metastatic melanoma
* Adequate hematological, renal, and liver function
* Negative serum pregnancy test at screening
* Fertile men and women must use an effective form of contraception during the study and for at least 6 months after completion of the study

Exclusion Criteria:

* Evidence of symptomatic CNS lesions as determined by the investigator, use of steroid or anti-seizure medication for treatment of brain metastases prior to the first administration of vemurafenib
* Patients with previous malignancies (other than melanoma) within the past 2 years except patients with treated and controlled basal or squamous cell carcinoma (SCC) of the skin or carcinoma in-situ of the cervix.
* Concurrent administration of any anti-cancer therapies (e.g. chemotherapy, other targeted therapy, experimental drug, etc.) other than those administered in this study
* Known hypersensitivity to vemurafenib or another BRAF inhibitor
* Pregnant or lactating women
* Refractory nausea and vomiting, malabsorption, external biliary shunt, or significant bowel resection that would preclude adequate absorption.
* Any of the following within the 6 months prior to the first vemurafenib administration: myocardial infarction, severe/unstable angina, symptomatic congestive heart failure, cerebrovascular accident or transient ischaemic attack, pulmonary embolism, hypertension not adequately controlled by current medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-10-17 (Actual); Primary Completion 2019-05-22 (Actual); Study Completion 2019-05-22 (Actual)

PRIMARY OUTCOMES:
Safety: Incidence of adverse events | 12 months

SECONDARY OUTCOMES:
Overall response rate according to Response evaluation criteria in solid tumors (RECIST v1.1) | 12 months
Progression free survival | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (9):
- South Africa (9):
  - National Hospital; Oncotherapy Dept, Bloemfontein
  - Groote Schuur Hospital ( Uni of Capetown ); Oncology Dept, Cape Town
  - Cape Town Oncology Trials, Cape Town
  - Cancercare, Cape Town
  - Cancercare, George
  - Mary Potter Oncology Centre, Groenkloof
  - Medical Oncology Centre of Rosebank; Oncology, Johannesburg
  - University of Pretoria; Department of Medical Oncology, Pretoria
  - Sandton Oncology Medical Group, Sandton